CLINICAL TRIAL: NCT06962930
Title: A Pilot RCT of a Remote Physical Activity Coaching Intervention to Promote Engagement in Physical Activity for People With Parkinson's Disease in Qatar
Brief Title: An Online Physical Activity Coaching Intervention for People With PD in Qatar
Acronym: EQP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qatar University (Other)
Collaborators: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Hanan Khalil, professor, Qatar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QU-CG/CHS-24/25-498; QU-IRB063/2024-EA (Other Grant/Funding Number: Qatar University)
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
Keywords: PD: Parkinson's Disease PA: Physical Activity NDD: Neuro Degenerative Disease QRI: Qatar Rehabilitation Institute
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): Participants will receive an 8-week personalized self-management program. They will be invited to one to 4 face-to-face coaching sessions and 7 remote online sessions. The first session will lay the groundwork for the program, in which an orientation of the features of the online forum will be provided. In addition, goal setting, use of smart watch to record progress, and how to track progress will be discussed. During the remote sessions, the participant and coach will work through informational modules of how to overcome barriers to exercise engagement and how to manage PD symptoms. The coach will provide encouragement in relation to regular physical activity and exercise, and the participant will report on progress related to goals they developed. All participants will receive a wearable watch to help them monitor their physical activity; although wearing the watch is optional, we will recommend that all participants wear it for the 12-week intervention.
  Interventions: Other: 8-week personalized self-management program tailored to their individual needs using Engage-Qatar PD. participants will be invited to one face-to-face coaching session and 7 online sessions
- Control group (Active Comparator): Participants in the control group will receive information on the published recommendations for physical activity for people with PD43. This is the standard information related to physical activity that an individual with PD would be expected to receive from their healthcare provider. To control for the ubiquitous nature of technology, all control participants will also receive Fitbit watches with basic instructions for monitoring their levels of physical activity. As in the intervention group, use of the Fitbit is optional, though we will recommend that both groups wear it for the 8-week intervention. The key ingredients of Engage-Qatar PD are the personalized coaching and self-management approach; thus, the control group will not have access to the Engage-Qatar PD online forum, nor will they have access to coaching or any component of the self-management approach.
  Interventions: Other: 8-week personalized self-management program tailored to their individual needs using Engage-Qatar PD. participants will be invited to one face-to-face coaching session and 7 online sessions

INTERVENTIONS:
Other: 8-week personalized self-management program tailored to their individual needs using Engage-Qatar PD. participants will be invited to one face-to-face coaching session and 7 online sessions — The first session will lay the groundwork for the program, in which an orientation of the features of the online forum will be provided. In addition, goal setting, use of watches, and how to track progress will be discussed. During the remote sessions, the participant and coach will work through informational modules of how to overcome barriers to exercise engagement and how to manage PD symptoms. In addition, the coach will provide encouragement in relation to regular physical activity and exercise, and the participant will report on progress related to up to three realistic and individualized goals they developed. key elements: (1) participant-therapist interaction, (2) online forum featuring a physical activity guidebook and workbook, (3) an online platform with personal physical activity database, (4) a wearable smart watch for activity monitors, (5) a video exercise library, (6) online support group, and (7) incorporate adaptation to Arabic culture and available in Arabic

SUMMARY:
Regular exercise can improve function and quality of life as well as have other positive behavioral and health-related benefits in people Parkinson's disease (PD). Despite the benefits, insufficient exercise is common among PD individuals, often due to common barriers, emphasizing the importance of empowering individuals with adequate knowledge and self-management skills.

This project aims to develop "Engage-Qatar PD," an online physical activity self-management program for people with PD in Qatar. Engage-Qatar PD will be grounded in a previously developed coaching intervention used in people with Huntington's disease (Engage HD) and people with PD. The main focus of this project will be the development work to adapt this intervention for online delivery for people with PD and within the Qatari context.

This development stage will entail participatory design, in which users will be actively involved as co-designers to ensure fully the required cultural adaptations. Following this development phase, a pilot randomized controlled trial will be conducted to assess the feasibility, acceptability, and potential benefits of the developed intervention.

The innovative approach proposed for this project would have wide-reaching impact, advancing the development of new therapeutic options. It will deliver a realistic, culturally adapted therapeutic option for people with PD in Qatar that has the potential to be implemented in a variety of healthcare settings and other countries in the region. Importantly, future work could replicate this program in a larger cohort of individuals with other neurodegenerative diseases and extend this work to other countries in the region.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years.
2. Successful completion of Physical Activity Readiness Questionnaire (PAR-Q), or medical clearance from a neurologist.
3. Ambulatory for indoor and outdoor mobility with or without an assistive device but without physical assistance.
4. A neurologist-confirmed diagnosis of PD.
5. Ability to follow study-related commands.

Exclusion Criteria:

1. Musculoskeletal injury or a medical condition that would prevent safe participation in an exercise program including failure to pass the PAR-Q test.
2. The presence of any other neurological conditions.
3. Acute illness or injury that prevents participation in the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Objective Physical activity | 7 days
  7 day physical activity (i.e., moderate/vigorous activity minutes) using a waist-worn activity monitor (Actigraph)

SECONDARY OUTCOMES:
The Physical Activity Scale for Individuals with Physical Disabilities (PASIPD) | less than 5 minutes
  Modified disability version of the 10 item Physical Activity Scale for the Elderly (PASE), Captures information about leisure, household, and work-related physical activity over the preceding 7 days, Developed targeting individuals with visual/auditory and locomotor/SCI disabilities.
International Physical Activity Questionnaire (IPAQ) short form | 5 minutes
  This measure will ask about the time spent being physically active in the last 7 days. The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity.
Six-Minute Walk Test (6MWT) | 10 minutes
  The 6-Minute Walk test is a measure of endurance. The Subjects will be asked to walk around the perimeter of a set circuit for a total of 6 minutes.
The Short Self-Efficacy for Exercise Scale (SSEE) | 5 minutes
  is a self-report questionnaire composed of nine items for the assessment of self-efficacy for exercise
8-item Parkinson's Disease Questionnaire (PDQ-8) | 5-10 minutes
  The 8-item version of the Parkinson's Disease Questionnaire (PDQ-8) is a shortened version of the 39-item Parkinson's Disease Questionnaire (PDQ-39). It was developed to reduce the respondent burden and increase convenience for use among persons with Parkinson's Disease in clinical settings. PDQ-39 comprises 39 questions from 8 dimensions which include mobility, activities of daily of living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort.PDQ-8 was constructed by taking one question from each domain of PDQ-39
MDS-UPDRS-II Motor Experiences of Daily Living | 10 minutes
  The unified Parkinson's disease rating scale (UPDRS) is used to follow the longitudinal course of Parkinson's disease. The UPD rating scale is the most commonly used scale in the clinical study of Parkinson's disease. . It is consisting of 4 parts one of them is MDS-UPDRS-II Motor Experiences of Daily Living it's about motor aspects of experiences of daily living (M-EDL).
MDS-UPDRS-III Motor Examination | 15 minutes
  The unified Parkinson's disease rating scale (UPDRS) is used to follow the longitudinal course of Parkinson's disease. The UPD rating scale is the most commonly used scale in the clinical study of Parkinson's disease. It is consists of 4 parts one of them is MDS-UPDRS-III Motor Examination its assesses the motor signs of PD
Levodopa Equivalent Daily Doses (LEDD) | 5 minutes
  The Levodopa Equivalent Daily Dose (LEDD) is a useful calculation for comparing the doses of different Parkinson's disease medications to their equivalent amount of Levodopa. This helps clinicians to evaluate the overall dopaminergic load a patient is receiving. Various Parkinson's medications, such as Levodopa, Dopamine Agonists, and MAO-B inhibitors, can be converted into an equivalent dose of Levodopa using standard conversion factors.
Mini Balance Evaluation Systems Test (Mini-BEST) | 10-15 minutes
  balance assessment tool is a shortened version of the Balance Evaluation Systems Test (BESTest) consists of 14 items, including 4 of the 6 sections (anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait) from the BESTest. It aims to target and identify 6 different balance control systems so that specific rehabilitation approaches can be designed for different balance deficits. The BESTest was shortened based on factor analysis to include dynamic balance only and to improve clinical utilization.
Five Times Sit to Stand Test (5TSTS) | Less than 5 minutes Depends on the number of trials
  The Five Times Sit to Stand Test measures one aspect of transfer skill. The test provides a method to quantify functional lower extremity strength and identify movement strategies a patient uses to complete transitional movements.
the Montréal Cognitive Assessment Scale (MOCA) | 10 minutes
  (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, vasoconstrictional skills, conceptual thinking, calculations, and orientation. The MoCA may be administered by anyone who understands and follows the instructions
the Symbol Digit Modalities Test | less than 5 minutes
  a commonly used test to assess psychomotor speed, which measures processing speed as well as motor speed. requires an individual to substitute digits for abstract symbols using a reference key. Performance is also affected by attention, visual scanning and tracking, and working memory .The SDMT has excellent psychometric properties, with high reliability and validity .
the Stroop Color-Word Interference | 5 minutes
  The Stroop Test is a measure of working memory and attention. When the colours and words a conflicting, the brain must work hard to filter out competing signals. Reading is such an automatic task that the brain needs to actively inhibit it and direct its attention instead to saying the colour of the letters. The resulting delay is called the Stroop Effect. When the colours and words match, or when the words are neutral, there is no conflicting information for the brain to have to filter out.
Pittsburgh sleep quality index (PSQI) | 5-10 minutes
  is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score It is a valuable tool for assessing sleep quality as it captures multiple dimensions of sleep, including both subjective experiences and objective parameters. It allows researchers and healthcare providers alike to obtain a comprehensive understanding of an individual's sleep patterns and disturbances.
the Hospital Anxiety-Depression scale (HADS) | 2-5 minutes
  is a 14-item scale, with seven items relating to anxiety and seven relating to depression.
10 Meter Walk Test (10MWT) | 5 minutes
  The 10 Meter Walking Test (10 MWT) assesses short duration walking speed (m/s). It has been used various patient populations including stroke, Parkinson's disease and general neurologic movement disorders.
  The 10 Meter Walking Test (10 MWT) is clinician-administered, and measures the time required to walk 10 meters. The test is performed using a "flying start": the patient walks 14m, and the time is measured for the intermediate 10 meters.
Barriers to Being Active Quiz (BBAQ) | 5-10 minutes
  is a structured questionnaire that measures the barriers to being active consists of 21 questions.
Barriers Subscale of the Physical Fitness | 5-10 minutes
  It a 21-item measure assessing the following barriers to physical activity: 1) lack of time, 2) social influence, 3) lack of energy, 4) lack of willpower, 5) fear of injury, 6) lack of skill, and 7) lack of resources. Each domain contains 3 items, with a total score range of 0 to 63. Respondents rate the degree of activity interference on a 4-point scale, ranging from 0 = "very unlikely" to 3 = "very likely."
The Modified Fatigue Impact Scale | 5-10 minutes
  self-report questionnaire provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning and it consists of 21 items.
Barriers to Health Promoting Activities for Disabled Persons Scale (BHADP) | 5-10 min
  an 18-item, 4-point scale to measure individual barriers to taking care of health. The original scale had 16 items; two additional barrier items, these items address the weather and lack of help from health care professionals. Respondents are asked to indicate how often listed barriers keep them from taking care of their health. Items include intrapersonal, interpersonal, and environmental barriers. Examples of barriers include being too tired, having other responsibilities, and lack of transportation.
7 day physical activity (i.e., step count) using a waist-worn activity monitor (Actigraph) | 7 days

CONTACTS AND LOCATIONS:
Locations (3):
- Qatar (3):
  - Qatar Rehabilitation Institution, Doha
  - Rumaila Hospital, Doha
  - Qatar University, Doha

IPD SHARING:
Plan to Share IPD: No